CLINICAL TRIAL: NCT00420381
Title: A Phase II Evaluation of Enzastaurin in the Treatment of Persistent or Recurrent Ovarian or Primary Peritoneal Carcinoma
Brief Title: Evaluation of Enzastaurin in the Treatment of Persistent or Recurrent Ovarian or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10738; H6Q-MC-S025 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-01-08; First posted 2007-01-11 (Estimated); Results first posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-11

CONDITIONS: Ovarian Cancer; Neoplasms; Carcinoma
Keywords: Recurrent Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms; Carcinoma; Recurrence | interventions — enzastaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Drug: enzastaurin

INTERVENTIONS:
Drug: enzastaurin — 1125 mg loading dose then 500 mg, oral, daily, until progressive disease
  Other Names: LY317615

SUMMARY:
The purpose is to assess the efficacy and toxicity of the study agent, enzastaurin, in participants with recurrent or persistent ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have recurrent or persistent epithelial ovarian or primary peritoneal carcinoma.
* All participants must have measurable disease.
* Participants must have at least one "target lesion" to be used to assess response on this protocol.
* Participants must not be eligible for a higher priority GOG protocol, if one exists.
* Participants who have received one prior regimen must have a GOG Performance Status of 0, 1, or 2. Participants who have received two prior regimens must have a GOG Performance Status of 0 or 1.
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration. Continuation of hormone replacement therapy is permitted.
* Any other prior therapy directed at the malignant tumor, including immunologic agents, must be discontinued at least four weeks prior to registration.
* Participants must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound.
* Participants must NOT have received any non-cytotoxic therapy for management of recurrent or persistent disease.
* Participants of child-bearing potential must have a negative serum pregnancy test prior to study entry and be practicing an effective form of contraception (for example, intrauterine device [IUD], birth control pills, or barrier device) during and for 3 months after discontinuation of study treatment.

Exclusion Criteria:

* Participants with previous enzastaurin treatment.
* Participants who have received radiation to more than 25% of marrow-bearing areas
* Participants with other invasive malignancies, with the exception of non-melanoma skin cancer, who had (or have) any evidence of other cancer present within the last 5 years or whose previous cancer treatment contraindicates this protocol therapy.
* Participants who have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Participants who are unable to discontinue use of carbamazepine, phenobarbital, and phenytoin (refer to Concomitant Medications for a discussion of enzyme inducing anti-epileptic drugs [EIAEDs]).
* Participants who are receiving concurrent administration of any other systemic anticancer therapy except for a biphosphonate if patient has bony metastases.
* Participants who have received prior therapy with non-cytotoxic agents (i.e. bevacizumab).
* Participants with serious concomitant systemic disorders (for example, active infection or abnormal electrocardiogram (ECG) indicative of cardiac disease) that, in the opinion of the investigator, would compromise the safety of the patient and his/her ability to complete the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Usha, Study Director — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group 215-854-0770, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers are defined as receiving at least one dose of study drug and treated until progressive disease.
Groups:
- Enzastaurin: 1125 mg oral loading dose enzastaurin then 500 mg, oral, daily, until progressive disease.
Period: Overall Study
Arm/Group | Enzastaurin
Started | 28
Received at Least One Dose of Study Drug | 27
Completed | 27
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Arm/Group | Enzastaurin
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival for at Least 6 Months (PFS-6)
Description: Data presented are the percentage of participants without progressive disease (PD) or death from any cause 6 months after registration. PD was a 25% increase in the sum of products of all measurable lesions (or 2 largest lesions if too numerous) over the smallest sum observed (over baseline if no decrease) or clear worsening of any evaluable disease, or appearance of any new lesion/site, or failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: Baseline through 6 months
Population: All participants who received at least 1 dose of study drug. 1 participant was censored.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 26
Percentage of participants | 10 [0 to 20]

2. Primary Outcome: Number of Participants With Adverse Events and Severe Adverse Events
Description: Data presented are the number of participants who experienced 1 or more adverse events (AEs) (all causalities and drug-related) and serious AEs (SAEs). A summary of SAEs and other non-serious AEs, regardless of causality is located in the Reported Adverse Events section of this record.
Time Frame: Baseline through end of study (Up to 45 months)
Population: All enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 28
Participants
  Other AEs | 27
  SAEs | 12

3. Secondary Outcome: Duration of Progression-Free Survival
Description: PFS is defined as the rate of PFS from the date of diagnosis to the first date of objectively determined progressive disease (based on radiological assessment) or death from any cause. It is assumed that PFS follows an exponential distribution.
Time Frame: Baseline to disease progression (Up to 38 months)
Population: All participants who received at least 1 dose of study drug, 1 participant was censored.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Enzastaurin
Number analyzed (Participants) | 26
months | 1.9 [1.5 to 2.7]

4. Secondary Outcome: Prognostic Factors: Platinum Sensitivity
Description: Participants who had disease progression within 6 months of ending their last regimen of platinum therapy were considered platinum resistant. Participants who had disease progression between 6 and 12 months of ending their last platinum regimen were considered platinum sensitive. Participants who had disease progression beyond 12 months of ending their last platinum regimen were also considered platinum sensitive.
Time Frame: Baseline
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 27
Participants
  Refractory Resistant (<6 months) | 17
  Sensitive (>= 6months) | 9
  Missing | 1

5. Secondary Outcome: Prognostic Factors: Performance Status
Description: Performance Status 0 = Fully active, able to carry on all pre-disease performance without restriction Performance Status 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature, e.g., light housework, office work.
Time Frame: Baseline
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin
Number analyzed (Participants) | 27
Participants
  Performance Status 0 | 16
  Performance Status 1 | 11

6. Secondary Outcome: Overall Survival
Description: Overall survival (OS) time is defined as the time from the date of diagnosis to the date of death from any cause. For participants who are still alive at the time of analysis, survival time will be censored at the last contact date.
Time Frame: Baseline through end of study (Up to 45 months)
Population: All participants who received at least one dose of study drug. 8 participants were censored.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Enzastaurin
Number analyzed (Participants) | 19
Months | 15.1 [9.5 to 33.3]

ADVERSE EVENTS:
Description: All participants in study.
Arm/Group | Enzastaurin
Serious Adverse Events (participants affected / at risk) | 12/28
Other Adverse Events (participants affected / at risk) | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin (N=28)
Hypertension (Cardiac disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (3)
Insomnia (General disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)
Death not associated with ctcae term (General disorders) | 3 (3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (2)
Ascites (non-malignant) (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (3)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (2)
Gastrointestinal - other (Ascites Malignant) (Gastrointestinal disorders) | 1 (1)
Ileus, gi (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1 (1)
Incontinence, anal (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Obstruction, gi (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (5)
Hemorrhage, gi (Blood and lymphatic system disorders) | 2 (2)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Blood and lymphatic system disorders) | 1 (1)
Edema: limb (General disorders) | 1 (2)
Creatinine (Metabolism and nutrition disorders) | 1 (2)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Pain (General disorders) | 4 (7)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Pulmonary/upper respiratory - other (Malignant Pleural Effusion) (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin (N=28)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 4 (9)
Allergy/immunology - other (Immune system disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 16 (35)
Insomnia (General disorders) | 2 (2)
Sweating (diaphoresis) (General disorders) | 2 (2)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 2 (3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (9)
Anorexia (Gastrointestinal disorders) | 10 (16)
Ascites (non-malignant) (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 9 (18)
Diarrhea (Gastrointestinal disorders) | 13 (20)
Distension/bloating, abdominal (Gastrointestinal disorders) | 2 (2)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 3 (3)
Heartburn/dyspepsia (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 10 (23)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (6)
Infection with normal anc or grade 1 or 2 neutrophils (Infections and infestations) | 6 (30)
Edema: limb (General disorders) | 6 (9)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3 (5)
Alkaline phosphatase (Metabolism and nutrition disorders) | 3 (4)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (2)
Creatinine (Metabolism and nutrition disorders) | 2 (2)
Glomerular filtration rate (Metabolism and nutrition disorders) | 3 (4)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 3 (6)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 (3)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (2)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (3)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 4 (8)
Mood alteration (General disorders) | 2 (3)
Pain (General disorders) | 17 (32)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Urine color change (Renal and urinary disorders) | 3 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days